CLINICAL TRIAL: NCT00261352
Title: A 24-Week Randomised, Double-Blind, Parallel-Group, Multi-Centre, Active-Controlled (Metformin or Metformin Combined With Fenofibrate) Study to Evaluate the Lipid Metabolic Effects, Safety and Tolerability of Tesaglitazar Therapy in Patients With Type 2 Diabetes and Low HDL-Cholesterol on a Fixed Background Therapy With a Statin
Brief Title: GALLANT 14 Tesaglitazar vs. Metformin and Fenofibrate
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C00003; EudraCT No 2004-02550-56
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar; Metformin; Fenofibrate

INTERVENTIONS:
Drug: Tesaglitazar
Drug: Metformin
Drug: Fenofibrate

SUMMARY:
This is a 24-week study to determine the lipid metabolic effects, safety, and tolerability of tesaglitazar compared with metformin and metformin in combination with fenofibrate in patients with type 2 diabetes and low high-density lipoprotein cholesterol (HDL-C). Improvement in dyslipidemia will be evaluated. The study comprises a 2-week enrollment period, 6-week run-in and a 24-week randomized, double blind, parallel group, multi-center, active controlled (metformin with or without fenofibrate) treatment period and a 3-week follow-up. From visit 2 (run-in), all patients will receive a standardized dose of statin (rosuvastatin)

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >=18 years of age
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Diagnosed with type 2 diabetes
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral antidiabetic agents

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above the normal range
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2005-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The change in HDL-C from baseline to the end of the randomized treatment period.

SECONDARY OUTCOMES:
Changes in the following variables from baseline to the end of the randomized treatment period:
Lipid and lipoprotein variables (triglycerides [TG], non-HDL-C, total cholesterol, low-density lipoprotein cholesterol [LDL-C], lipoprotein particle size and concentration, free fatty acid, apolipoprotein [Apo] AI, Apo B, Apo CIII)
Responder analyses for HDL-C, TG, and non-HDL-C according to pre-specified values
The proportion of patients reaching pre-specified target levels for HDL-C, TG, and non-HDL-C
Risk markers for cardiovascular disease (C-reactive protein, insulin, homeostasis model assessment, LDL-C/HDL-C ratio, very-low-density lipoprotein cholesterol/LDL-C ratio, Apo B/Apo AI ratio)
Central obesity (waist/hip ratio)
Pharmacokinetics of tesaglitazar
Safety and tolerability of tesaglitazar by assessment of adverse events, laboratory values, electrocardiogram, pulse, blood pressure, hypoglycemic events, body weight, cardiac evaluation, and physical examination

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science DIrector, MD, Study Director — AstraZeneca
Locations (152):
- Brazil (5):
  - Research Site, Fortaleza, Ceará
  - Research Site, Goiânia, Goiás
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo
  - Research Site, Curitiba
- Canada (19):
  - Research Site, Calgary, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Bolton, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Hastings, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Napanee, Ontario
  - Research Site, Newboro, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Sherbrooke, Quebec
- Finland (12):
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Mikkeli
  - Research Site, Oulu
  - Research Site, Porvoo
  - Research Site, Savonlinna
  - Research Site, Seinäjoki
  - Research Site, Suonenjoki
  - Research Site, Tampere
  - Research Site, Turku
  - Research Site, Vaasa
- France (38):
  - Research Site, Aix-en-Provence
  - Research Site, Ambriere LES Vallees
  - Research Site, Béziers
  - Research Site, Briey
  - Research Site, Broglie
  - Research Site, Château-Gontier
  - Research Site, Cremeaux
  - Research Site, Falaise
  - Research Site, Fontaine Saint Martin
  - Research Site, Freyming-Merlebach
  - Research Site, Gan
  - Research Site, Hyères
  - Research Site, Jarny
  - Research Site, Jort
  - Research Site, L'Aigle
  - Research Site, Lambersart
  - Research Site, Le Lavandou
  - Research Site, Lille
  - Research Site, Lomme
  - Research Site, Marange-Silvange
  - Research Site, Marignane
  - Research Site, Mars-la-Tour
  - Research Site, Martigues
  - Research Site, Mayenne
  - Research Site, Metz
  - Research Site, Mondelange
  - Research Site, Montbrison
  - Research Site, Montpellier
  - Research Site, Moûtiers
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Roanne
  - Research Site, Roquevaire
  - Research Site, Rugles
  - Research Site, Saint-Chamond
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Tantonville
- Germany (22):
  - Research Site, Heidelberg, Baden-Wurttemberg
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, München, Bavaria
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Hanover, Lower Saxony
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Dresden, Saxony
  - Research Site, Berlin, State of Berlin
  - Research Site, Aschaffenburg
  - Research Site, Beckum
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Gelnhausen
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Künzing
  - Research Site, Nuremberg
  - Research Site, Pirna
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Hungary (8):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Gy¿r
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Siófok
  - Research Site, Székesfehérvár
- India (4):
  - Research Site, Mumbai, Mashatra
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, India
- Indonesia (2):
  - Research Site, Jakarta, DKI Jakarta
  - Research Site, Malang, East Java
- Malaysia (3):
  - Research Site, George Town
  - Research Site, Kuala Lumpur
  - Research Site, Petaling Jaya
- Norway (9):
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Elverum
  - Research Site, Fredrikstad
  - Research Site, Hamar
  - Research Site, Oslo
  - Research Site, Paradis
  - Research Site, Trondheim
  - Research Site, Tvedestrand
- Philippines (3):
  - Research Site, Cebu City
  - Research Site, Makati City
  - Research Site, Manila
- Portugal (6):
  - Research Site, Almada
  - Research Site, Amadora
  - Research Site, Caldas da Rainha
  - Research Site, Elvas
  - Research Site, Lisbon
  - Research Site, Portalegre
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Research Site, Singapore, Singapore
- South Africa (4):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Pretoria
- Switzerland (7):
  - Research Site, Bern
  - Research Site, Chur
  - Research Site, Ilanz
  - Research Site, Lausanne
  - Research Site, Monthey
  - Research Site, Sion
  - Research Site, Zurich
- Taiwan (4):
  - Research Site, Yongkang District, Tainan County
  - Research Site, Changhua
  - Research Site, Taichung
  - Research Site, Taipei